CLINICAL TRIAL: NCT03227328
Title: Group Sequential Response Adaptive Randomized Clinical Trial of Concomitant Chemotherapy Plus Endocrine Therapy Versus Cyclin-dependent Kinase 4/6 (CDK4/6) Inhibitor Plus Endocrine Therapy for Advanced Hormone Receptor-positive, HER2-negative Breast Cancer.
Brief Title: CDK4/6-inhibitor or Chemotherapy, in Combination with ENDOcrine Therapy, for Advanced Breast Cancer / KENDO
Acronym: KENDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.19; 2016-004107-31 (EudraCT Number)
Record Dates: First submitted 2017-07-19; First posted 2017-07-24 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Hormone Receptor Positive Breast Cancer; Metastatic Breast Cancer; Hormone Receptor Negative Breast Cancer
Keywords: HR-positive Breast Cancer; metastatic breast cancer; First line treatment; endocrine therapy; chemotherapy; randomized phase III trial; aromatase inhibitor; HR-negative Breast Cancer; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: group sequential response adaptive Randomized, open label, multicenter,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm A (Active Comparator): concomitant cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor plus endocrine therapy
  Interventions: Drug: concomitant cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor plus endocrine therapy
- Treatment Arm B (Experimental): chemotherapy plus endocrine therapy (administered either concomitantly or sequentially)
  Interventions: Drug: chemotherapy plus endocrine therapy (administered either concomitantly or sequentially)

INTERVENTIONS:
Drug: concomitant cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor plus endocrine therapy — CDK4/6 inhibitor:
  * palbociclib
  * ribociclib
  * abemaciclib
  Endocrine therapy:
  * non-steroidal or steroidal AI
  * fulvestrant
  Arms: Treatment Arm A
Drug: chemotherapy plus endocrine therapy (administered either concomitantly or sequentially) — Standard Chemotherapy regimens will be classified as:
  * anthracycline + taxane,
  * taxane,
  * anthracycline,
  * capecitabine / fluoropyrimidines,
  * others.
  Endocrine therapy:
  * non-steroidal or steroidal AI
  * fulvestrant
  Arms: Treatment Arm B

SUMMARY:
Prospective, open label, multicenter, group sequential response adaptive randomized phase 2 study, comparing two treatments for locally advanced or metastatic luminal breast cancer:

* Arm A: concomitant cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor (palbociclib, ribociclib or abemaciclib) plus endocrine therapy (aromatase inhibitor [AI] or fulvestrant)
* Arm B: chemotherapy plus endocrine therapy (AI or fulvestrant, administered either concomitantly from the beginning of chemotherapy or sequentially after 4-6 months of chemotherapy) Treatments will continue until disease progression or toxicity or patient refusal.

DETAILED DESCRIPTION:
Group sequential response adaptive randomized clinical trial of concomitant chemotherapy plus endocrine therapy versus cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor plus endocrine therapy for advanced hormone receptor-positive, HER2-negative breast cancer Primary Objective: To compare the efficacy of concomitant CDK4/6 inhibitor plus endocrine therapy versus chemotherapy plus endocrine therapy (administered either concomitantly from the beginning or sequentially) in terms of progression-free survival (PFS).

Secondary objectives: To compare between treatment arms:

* quality of life (EORTC quality of life questionnaire(QLQ) QLQ -C30 and QLQ-BR23)
* toxicity (CTCAE version 5.0)
* time to treatment failure
* best response rate
* duration of response
* clinical benefit rate
* overall survival (OS)
* PFS and clinical benefit with the subsequent line of treatment after cross-over: CDK4/6 inhibitors plus endocrine therapy in patients treated with chemotherapy plus endocrine therapy, chemotherapy (with or without endocrine therapy) in patients treated with CDK4/6 inhibitors plus endocrine therapy
* correlative biomarkers of response to CDK4/6 inhibitors and chemotherapy:

  * tissue markers (on the primary tumor and / or metastatic tissue)
  * circulating markers (e.g. CTCs, ctDNA)

The patients will be allocated according to block randomization until two events are observed in each arm, and then according to the time-to-event adaptation of the group sequential Doubly-adaptive Biased Coin Design (DBCD) whose allocation probabilities are computed at the end of the block randomization and after around 70% and 85% of the 150 maximum patients are enrolled during a 23 month period. At these last two (i.e. after 105 and 128 patients, respectively), interim analysis on efficacy will be carried out allowing for early stopping. At the end of the 16-month follow up, administrative censoring is introduced. Therefore, the total study duration is 39 months.

Previous results on palbociclib and fulvestrant combination in second line and the characteristics of our target population lead us to assume a median PFS of 8 and 12 months for arm A and B, respectively. Under this scenario, for a sample size of at the most 150 patients, the proposed design strategy has led to a simulated power of 0.911 compared with a 0.717 one for the Complete Randomisation design.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of HR-positive (ER ≥10% of tumor cells), HER2-negative breast cancer, determined by local laboratory on most recent available tumor tissue.
* Locally advanced (not susceptible to locoregional therapy) or metastatic disease (herein globally defined as "advanced breast cancer (ABC)").
* At least one of the following signs of disease aggressiveness:

  * The main criteria are a low expression of ER (10% ≤ ER < 50%) and/or a relapse while on the first 2 years of adjuvant endocrine therapy or disease progression (PD) within the first 6 months of first-line endocrine therapy for ABC
  * Other tumor characteristics of aggressiveness that make the patient potentially candidate to chemotherapy, according to the guidelines of the Italian Association of Medical Oncology [AIOM guidelines 2017], such as: elevated Ki67 (preferably documented, if available, on a metastatic biopsy), low expression of hormone receptors (e.g. progesterone receptor <20%), extended visceral involvement or visceral involvement at risk for organ failure, uncontrolled symptoms; these patients are eligible if chemotherapy is considered a suitable option by the treating physician.
* Postmenopausal women, or premenopausal women undergoing treatment with LHRH analog, or men (either receiving treatment with LHRH analog or not).
* Measurable disease according to RECIST 1.1 criteria, or not measurable but evaluable disease.
* Any prior adjuvant chemotherapy or endocrine therapy
* No prior chemotherapy for advanced disease.
* Up to one prior line of endocrine therapy for ABC.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group performance status (ECOG-PS) ≤2 (see Appendix A).
* Adequate organ (renal, hepatic, bone marrow, cardiac) functions.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to use effective contraception during the study period and for 4 months thereafter. Effective contraception methods include: total abstinence (when this is in line with the preferred and usual lifestyle of the subject); tubal ligation; male sterilization; combination of the placement of an intrauterine device or intrauterine system and barrier methods of contraception with spermicidal suppository.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Any prior chemotherapy or CDK4/6 inhibitor for advanced breast cancer
* More than 1 prior line of endocrine therapy for ABC.
* Patients who have not recovered from adverse events due to prior therapies to grade ≤1 (excluding alopecia).
* Active central nervous system metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the drugs used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior history of non-breast malignancy (except for adequately controlled basal cell carcinoma of the skin, carcinoma in situ of the cervix, in situ carcinoma of the bladder), unless treated with curative intent and disease free for at least 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 39 months
  time from randomization until first disease progression or death; disease progression is defined according to Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1

SECONDARY OUTCOMES:
EORTC QLQ-C30 quality of life between the 2 arms | up to 39 months
  evaluation of EORTC QLQ-C30 Version 3.0
QLQ-BR23 quality of life between the 2 arms | up to 39 months
  evaluation of QLQ-BR23 (breast cancer specific)
toxicity | up to 39 months
  evaluation of toxicity by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
time to treatment failure (TTF) | up to 39 months
  the time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient refuse or death.
best objective response rate | up to 39 months
  best objective (partial or complete) response rate according to RECIST 1.1
duration of response | up to 39 months
  time from documentation of tumor response to disease progression
clinical benefit rate (CBR) | up to 39months
  the percentage of patients who achieved complete response, partial response or stable disease lasting longer than 24 weeks
overall survival (OS) | up to 39 months
  time from randomization until death for any cause
Progression free survival (PFS) | up to 39 months
  PFS and clinical benefit with the subsequent line of treatment after cross-overtime calculated from randomization until the date of start of the subsequent treatment line
correlative biomarkers of response to chemotherapy and endocrine therapy | up to 39 months
  correlative biomarkers assessed on baseline tumor specimens (from primary tumor or metastatic biopsies) and blood samples collected at baseline and at different timepoints until evidence of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rocca, Study Director — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Via Maroncelli 40, 47014 Meldola, ITALY
Locations (20):
- Italy (20):
  - U.O. Oncologia Medica, P.O. Bellaria-Maggiore, Bologna, BO
  - UO Oncologia Medica IRST IRCCS, Meldola, FC
  - Dip. Medicina Interna e Riabilitazione - U.O. Medicina Interna Oncologica, Ospedale Ramazzini, Carpi, MO
  - Dip. Oncologia-Ematologia - U.O. Oncologia Medica,Azienda USL di Piacenza - Ospedale Civile, Piacenza, PC
  - UOC Oncologia Medica AUSL Romagna-Ravenna, Ravenna, RA
  - UO Oncologia Medica AUSL Romagna-Rimini, Rimini, RI
  - A.O.U. Ospedali Riuniti Umberto I - GM Lancisi - G Salesi, Ancona
  - U.O. Oncologia Medica; Ist. Tumori Giovanni Paolo II - IRCCS Osp. Oncologico di Bari, Bari
  - Terapia Molecolare e Farmaco Genomica, Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - A.O.U. di Ferrara Arcispedale Sant'Anna, Ferrara
  - Ospedale Civile di Guastalla - AUSL di Reggio Emilia, Guastalla
  - AUSL Imola, Imola
  - Ospedale Mater Salutis - Azienda ULSS9 Scaligera, Legnago
  - Ospedale di Macerata, ASUR AV3, Macerata
  - A.O.U. Policlinico di Modena, Modena
  - A.O.U. Maggiore della Carità di Novara, Novara
  - U.O. Oncologia Medica, AOU di Parma, Parma
  - A.O. Santa Maria della Misericordia di Perugia, Perugia
  - A.O. Arcispedale S. Maria Nuova IRCCS di Reggio Emilia, Reggio Emilia
  - Ospedale di Sondrio - ASST Valtellina e Alto Lario, Sondrio